CLINICAL TRIAL: NCT04537039
Title: Prospective, Multicentric Study, Aiming to Assess the Relevance of a Frailty Screening by Home Care Services
Brief Title: Home Care Services Screening for Frailty.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID outbreak did not allow home visits
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FRAILTY
Record Dates: First submitted 2020-07-30; First posted 2020-09-03 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All the participants. (Other): This study only includes 1 arm.
  Interventions: Diagnostic Test: Frailty screening for people over 65 living at home.

INTERVENTIONS:
Diagnostic Test: Frailty screening for people over 65 living at home. — The home care services will carry out the SEGA-A test.

SUMMARY:
An improvement in professional practices on the topic of frailty is desirable as much for ambulatory care teams (professionals in home care services) than for hospital care teams (medical and paramedical). Geriatric prevention, screening for frailty, are major challenges for the years to come and require involvement and a know-how.

The main hypothesis is that the screening of the frailty of the elderly, by the home care services is relevant and reliable, therefore making it possible to detect a state of frailty and organize preventive care at the earliest.

The objectives of this research work are:

* to demonstrate that the use of a questionnaire, simple and already validated for a medical use, can be administered by home care services with just as much relevance,
* to democratize the detection of frailty by demonstrating that home care services have an important role to play in terms of screening and therefore an equally important impact in terms of public health,
* to recall the importance of screening in medical practice, including for the elderly.

DETAILED DESCRIPTION:
The continued increase in life expectancy is one of the most significant achievements of these years in Europe: while in 1960 life expectancy was 73.6 years for women and 67 years for men, in 2010 it was significantly higher, respectively 84.8 years and 78.1 years. Total life expectancy is increasing, but disability-free life expectancy is declining.

Thus, the years of life gained would now be accompanied by functional limitations, activity restrictions and degradation of autonomy. One of the challenges of our society, promoted as part of the European Innovation Partnership for Active and Healthy Aging as well as in the National Health Strategy 2018-2022, is the prevention of disabilities and age-related dependence by ensuring that our patients can not only live longer, but also lead a healthy, active and independent life.

The vast majority of older people live at home without significant disability, including in the most advanced age groups. These elderly pauci- or mono-pathological persons evolve in a manner comparable to younger adults in acute illness, hospitalization or during physical and / or psychological stress, the so-called "fragile" elderly unmask an underlying state of vulnerability and may enter into dependency.

In 2011, the French Society of Geriatrics and Gerontology (SFGG) adopted the following definition of frailty: "Frailty is a clinical syndrome. It reflects a decrease in physiological capacity reserve which alters the mechanisms of adaptation to stress. Its clinical expression is modulated by comorbidities and by psychological, social, economic and behavioral. Frailty syndrome is a marker of risk of mortality and pejorative events, including disabilities, falls, hospitalization and institutionalization. Age is a major determinant of frailty […]. Addressing the determinants of frailty can reduce or delay its consequences. Thus, fragility would be part of a process potentially reversible ".

According to the latest data from the SHARE survey (Survey on Health, Aging and Retirement in Europe) which is a multidisciplinary longitudinal Survey involving more than 80,000 Europeans aged over 50 with collection of data on health status, social situation (family, mutual aid, social networks) and economic (employment, retirement, wealth), frailty represents in France 3.2% of people aged 50 to 64, and 15% of people over 65. Other data of interest, 43% of people over 65 are "pre-fragile".

Thus, being able to identify fragility early is a major issue in order to implement corrective actions and avoid or at least delay entry into addiction. To do so, several simple primary care screening tools have been developed, like self-assessment such as the FiND8 self-questionnaire or tools intended to be used by physicians such as the FRAIL tool from Morley or the tool for identifying the frailty of the gerontopole of Toulouse.

These screening strategies remain mainly for the time in the medical field while home care services (SAD), daily actors in the elderly person life, are still too little involved. The development of Home Care Frailty Scale, a 29-item multidimensional assessment tool for the risk of decline to dependency, based on data from the interRAI (Resident Assessment Instrument), however, demonstrates that SAD represent an interesting screening strategy.

ELIGIBILITY:
Inclusion Criteria:

* Living at home.
* Functional independence preserved (ADL ≥ 5/6).
* Intervention of a Home Assistance Service (SAAD, SSIAD, carer, liberal nurse at home, etc.) for any reason.
* Signature of informed consent for the participation to the study.
* Affiliation to a social security scheme or beneficiaries of such a scheme.

Exclusion Criteria:

* Independency not preserved (ADL <5).
* Inability to understand the questions of the SEGA-A grid.
* Refusal to participate in the study expressed by the patient.
* Patients under guardianship or curatorship.
* Patient under end-of-life care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the performance of the SEGA-A test, used by professionals in the home care services, as a screening test for frailty of people over 65 living at home. | Date of the medical visit with the geriatrician.
  To measure the performance of the SEGA part A screening test (sensitivity, specificity, likelihood) used by the Home Care Services in screening for frailty, by comparing to the gold standard of the diagnosis of frailty represented by the Fried score, carried out by a doctor trained in geriatrics.
Evaluation of the performance of the SEGA-A test, used by professionals in the home care services, as a screening test for frailty of people over 65 living at home. | Date of the visit of the home care services.
  To measure the performance of the SEGA part A screening test (sensitivity, specificity, likelihood) used by the Home Care Services in screening for frailty, by comparing to the gold standard of the diagnosis of frailty represented by the Fried score, carried out by a doctor trained in geriatrics.

SECONDARY OUTCOMES:
To measure the feasibility of carrying out the screening test in current practice by home care services in terms of cost (financial and human) and acceptability. | Date of the visit of the home care services.
  To assess the feasibility of the screening test, the estimate duration of the SEGA-A grid will be measured in minutes.
To measure the feasibility of carrying out the screening test in current practice by home care services in terms of cost (financial and human) and acceptability. | Date of the visit of the home care services.
  To assess the feasibility of the screening test, the acceptability by the patient will be asked. This measurement will be given using a feasibility and acceptability questionnaire.
To measure the feasibility of carrying out the screening test in current practice by home care services in terms of cost (financial and human) and acceptability. | Date of the visit of the home care services.
  To assess the feasibility of the screening test, the acceptability by the professionnal will be filled in. This measurement will be given using a feasibility and acceptability questionnaire. This measurement will be done only once per professionnal regardless of the number of patients he took care of.
To evaluate the subjective feeling of the existence of frailty by home care services. | Date of the visit of the home care services.
  The subjective feeling of the state of frailty will be evaluated by the use of a numerical scale from 0 to 10, the score 0 corresponding to the perception of a robust state and the score 10 to that of a very fragile condition.
Epidemiology of the frailty of people in the care of the home care services and their relatives caregivers living at home (% robust, pre-fragile and fragile; to be done by age group). | Through study completion, an average of 2 years.
  The epidemiology of the frailty of people living at home for whom a home care service is involved will be calculated as a percentage and absolute value of robust, pre-fragile and fragile, according to the criteria determined by the Fried test.
To look for the elements associated with the diagnosis of frailty in order to have warning signs that should lead to a screening. | Through study completion, an average of 2 years.
  In order to find the guiding elements that would lead to screening of the frailty state, it will be a question of analyzing the correlation between the diagnosed state of frailty and the different medico-social data collected (medical background information).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique la chataigneraie, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morley JE, Malmstrom TK, Miller DK. A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging. 2012 Jul;16(7):601-8. doi: 10.1007/s12603-012-0084-2. PMID 22836700
- [Background] Vellas B, Balardy L, Gillette-Guyonnet S, Abellan Van Kan G, Ghisolfi-Marque A, Subra J, Bismuth S, Oustric S, Cesari M. Looking for frailty in community-dwelling older persons: the Gerontopole Frailty Screening Tool (GFST). J Nutr Health Aging. 2013 Jul;17(7):629-31. doi: 10.1007/s12603-013-0363-6. PMID 23933875
- [Background] Rolland Y, Benetos A, Gentric A, Ankri J, Blanchard F, Bonnefoy M, de Decker L, Ferry M, Gonthier R, Hanon O, Jeandel C, Nourhashemi F, Perret-Guillaume C, Retornaz F, Bouvier H, Ruault G, Berrut G. [Frailty in older population: a brief position paper from the French society of geriatrics and gerontology]. Geriatr Psychol Neuropsychiatr Vieil. 2011 Dec;9(4):387-90. doi: 10.1684/pnv.2011.0311. French. PMID 22182814
- [Background] Borsch-Supan A, Brandt M, Hunkler C, Kneip T, Korbmacher J, Malter F, Schaan B, Stuck S, Zuber S; SHARE Central Coordination Team. Data Resource Profile: the Survey of Health, Ageing and Retirement in Europe (SHARE). Int J Epidemiol. 2013 Aug;42(4):992-1001. doi: 10.1093/ije/dyt088. Epub 2013 Jun 18. PMID 23778574
- [Background] Vellas B, Cestac P, Moley JE. Implementing frailty into clinical practice: we cannot wait. J Nutr Health Aging. 2012 Jul;16(7):599-600. doi: 10.1007/s12603-012-0096-y. No abstract available. PMID 22836699
- [Background] Cesari M, Demougeot L, Boccalon H, Guyonnet S, Abellan Van Kan G, Vellas B, Andrieu S. A self-reported screening tool for detecting community-dwelling older persons with frailty syndrome in the absence of mobility disability: the FiND questionnaire. PLoS One. 2014 Jul 7;9(7):e101745. doi: 10.1371/journal.pone.0101745. eCollection 2014. PMID 24999805
- [Background] Morris JN, Howard EP, Steel KR. Development of the interRAI home care frailty scale. BMC Geriatr. 2016 Nov 21;16(1):188. doi: 10.1186/s12877-016-0364-5. PMID 27871235
- [Background] Sieliwonczyk E, Perkisas S, Vandewoude M. Frailty indexes, screening instruments and their application in Belgian primary care. Acta Clin Belg. 2014 Aug;69(4):233-9. doi: 10.1179/2295333714Y.0000000027. Epub 2014 Apr 29. PMID 24773077
- [Background] Zulfiqar AA. Identification of frailty by the use of the SEGAm scale (part A) in geriatrical consultation. Geriatr Psychol Neuropsychiatr Vieil. 2018 Sep 1;16(3):269-277. doi: 10.1684/pnv.2018.0740. PMID 29976541
- [Background] Oubaya N, Drame M, Novella JL, Quignard E, Cunin C, Jolly D, Mahmoudi R. Screening for frailty in community-dwelling elderly subjects: Predictive validity of the modified SEGA instrument. Arch Gerontol Geriatr. 2017 Nov;73:177-181. doi: 10.1016/j.archger.2017.07.026. Epub 2017 Aug 4. PMID 28822918
- [Background] Feck E, Zulfiqar AA. [Screening of frailty in family practice by the modified SEGA grid]. Rev Med Liege. 2018 Oct;73(10):513-518. French. PMID 30335257
- [Background] Tardieu E, Mahmoudi R, Novella JL, Oubaya N, Blanchard F, Jolly D, Drame M. [External validation of the short emergency geriatric assessment (SEGA) instrument on the SAFES cohort]. Geriatr Psychol Neuropsychiatr Vieil. 2016 Mar;14(1):49-55. doi: 10.1684/pnv.2016.0592. French. PMID 27005336
- [Background] Woo J, Yu R, Wong M, Yeung F, Wong M, Lum C. Frailty Screening in the Community Using the FRAIL Scale. J Am Med Dir Assoc. 2015 May 1;16(5):412-9. doi: 10.1016/j.jamda.2015.01.087. Epub 2015 Feb 24. PMID 25732832
- See also: Fiche de synthèse sur le questionnaire HS - F1109. — http://www.insee.fr/fr/publications-etservices/docs_doc_travail/F1109.pdf
- See also: Haute Autorité de Santé - Comment repérer la fragilité en soins ambulatoires ? — https://www.has-sante.fr/jcms/c_1602970/fr/comment-reperer-la-fragilite-en-soins-ambulatoires